CLINICAL TRIAL: NCT04883177
Title: Effectiveness and Safety of the COVID-19 Vaccination for Patients With Liver Disease (CHESS2101): a Multicenter Cohort Study
Brief Title: Effectiveness and Safety of the COVID-19 Vaccination for Patients With Liver Disease (CHESS2101)
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Huashan Hospital (Other); The Sixth People's Hospital of Shenyang City (Unknown); Xingtai City People's Hospital (Unknown); Jinchang Central Hospital (Unknown); Baoding People's Hospital (Unknown); The Third People's Hospital of Zhenjiang City (Unknown); Shanxi Bethune Hospital (Other); Wuhan Jinyintan Hospital (Unknown); Jincheng People's Hospital (Other); The Third People's Hospital of Tibet Autonomous Region (Unknown); People's Hospital of Ningxia Hui Autonomous Region (Other); Fuling Central Hospital of Chongqing City (Other); Hospital of the Chengdu Office of the People's Government of Tibet Autonomous Region (Unknown); The Central Hospital of Lishui City (Other); The Third People's Hospital of Linfen City (Unknown); Yibin First People's Hospital (Unknown); Jingzhou Central Hospital (Other); Wuxi Fifth People's Hospital (Unknown); Qingyang People's Hospital (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Beilun Hospital of Traditional Chinese Medicine (Unknown); Henan Provincial People's Hospital (Other); Qingdao Sixth People's Hospital (Unknown); The First Affiliated Hospital of Xiamen University (Other); Shandong Provincial Hospital (Other Government); Beijing YouAn Hospital (Other); The First People's Hospital of Taicang (Unknown); The Third People's Hospital of Taiyuan (Other); Tianjin Second People's Hospital (Other); Tianjin Third Central Hospital (Other); Qishan Hospital of Yantai City (Unknown); Affiliated Hospital of Yunnan University (Other); The First People's Hospital of Yunnan (Other); The Fourth Affiliated Hospital of Zhejiang University (Unknown); Third Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Chief, CHESS Center, Institute of Portal Hypertension, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2101
Record Dates: First submitted 2021-04-29; First posted 2021-05-12 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; Liver Disease; Vaccine Reaction
MeSH Terms: conditions — COVID-19; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 pandemic with SARS-CoV-2 infection has become a global challenge. Though most cases of COVID-19 are mild, the disease can also be fatal. Patients with liver disease are more susceptible to damage from SARS-CoV-2 infection considering their immunocompromised status. Therefore, early inoculation of SARS-CoV-2 vaccine in patients with liver disease is an important protective measure. However, information on the effectiveness and safety of the COVID-19 vaccine for liver disease remains to be determined. This muilticentre study (CHESS2101) aims to study the effectiveness and safety of the COVID-19 vaccination for patients with liver disease.

DETAILED DESCRIPTION:
Patients with liver disease, especially liver cirrhosis, hepatobiliary malignancies, candidates for liver transplantation, and individuals who are immunosuppressed after liver transplantation, have an increased risk of COVID-19 infection and increased mortality. Therefore, early inoculation of SARS-CoV-2 vaccine in liver disease patients is an important protective measure. A small number of SARS-CoV-2 vaccines have been tested in clinical trials in healthy individuals and have evidence of short-term safety, immunogenicity and efficacy. However, information on the effectiveness and safety of the COVID-19 vaccine for patients with liver disease remains to be determined. This muilticentre study (CHESS2101) aims to study the effectiveness and safety of the COVID-19 vaccination for patients with liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically or pathologically diagnosed with pre-existing liver disease, including: chronic liver disease, cirrhosis, liver cancer, liver transplant subjects, etc.;
2. Receiving the whole-course COVID-19 vaccination for 14 days or more;
3. Volunteer to participate in this study.

Exclusion Criteria:

1. Younger than 18 years old;
2. Women during pregnancy or lactation;
3. Research on other situations deemed unsuitable for selection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Populations With Liver Disease who Complete the whole-course COVID-19 vaccination
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events within 7 days after each injection | up to 7 days after each injection

SECONDARY OUTCOMES:
Overall incidence of adverse reactions within 28 days as assessed by CTCAE v4.0 | up to 28 days after each injection
Antibody serological conversion rate in populations with liver disease after COVID-19 vaccination | the day of the first dose of vaccination (baseline) and 14 days, 28 days, 90 days, and 180 days after the second dose of vaccination
Neutralizing antibody titers in blood samples after vaccination | the day of the first dose of vaccination (baseline) and 14 days, 28 days, 90 days, and 180 days after the second dose of vaccination
Antibody IgM titers in blood samples after vaccination | the day of the first dose of vaccination (baseline) and 14 days, 28 days, 90 days, and 180 days after the second dose of vaccination
Antibody IgG titers in blood samples after vaccination | the day of the first dose of vaccination (baseline) and 14 days, 28 days, 90 days, and 180 days after the second dose of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, MD, Study Chair — LanZhou University; Wenhong Zhang, MD, Study Chair — Huashan Hospital
Locations (37):
- China (37):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing You'an Hospital, Beijing, Beijing Municipality
  - Chongqing Fuling Central Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Jinchang Central Hospital, Jinchang, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Qingyang People's Hospital, Qingyang, Gansu
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - Baoding People's Hospital, Baoding, Heibei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Wuhan Jinyintan Hospital, Wuhan, Hubei
  - The First People's Hospital of Taicang, Taicang, Jiangsu
  - Wuxi Fifth People's Hospital, Wuxi, Jiangsu
  - The Affiliated Third Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qingdao Sixth People's Hospital, Qingdao, Shandong
  - Qishan Hospital of Yantai City, Yantai, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Jincheng People's Hospital, Jincheng, Shanxi
  - The Third People's Hospital of Linfen City, Linfen, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Taiyuan Third People's Hospital, Taiyuan, Shanxi
  - Hospital of the Chengdu Office of the People's Government of Tibet Autonomous Region, Chengdu, Sichuan
  - Yibin First People's Hospital, Yibin, Sichuan
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - The Third People's Hospital of Tibet Autonomous Region, Lhasa, Tibet
  - Affiliated Hospital of Yunnan University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Central Hospital of Lishui City, Lishui, Zhejiang
  - Beilun Hospital of Traditional Chinese Medicine, Ningbo, Zhejiang
  - The Fourth Affiliated Hospital of Zhejiang University, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] World Health Organization. Coronavirus disease (COVID-2019) situation reports[EB/OL]. https: //www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports/.
- [Background] Sarin SK, Choudhury A, Lau GK, Zheng MH, Ji D, Abd-Elsalam S, Hwang J, Qi X, Cua IH, Suh JI, Park JG, Putcharoen O, Kaewdech A, Piratvisuth T, Treeprasertsuk S, Park S, Wejnaruemarn S, Payawal DA, Baatarkhuu O, Ahn SH, Yeo CD, Alonzo UR, Chinbayar T, Loho IM, Yokosuka O, Jafri W, Tan S, Soo LI, Tanwandee T, Gani R, Anand L, Esmail ES, Khalaf M, Alam S, Lin CY, Chuang WL, Soin AS, Garg HK, Kalista K, Batsukh B, Purnomo HD, Dara VP, Rathi P, Al Mahtab M, Shukla A, Sharma MK, Omata M; APASL COVID Task Force, APASL COVID Liver Injury Spectrum Study (APCOLIS Study-NCT 04345640). Pre-existing liver disease is associated with poor outcome in patients with SARS CoV2 infection; The APCOLIS Study (APASL COVID-19 Liver Injury Spectrum Study). Hepatol Int. 2020 Sep;14(5):690-700. doi: 10.1007/s12072-020-10072-8. Epub 2020 Jul 4. PMID 32623632
- [Background] Iavarone M, D'Ambrosio R, Soria A, Triolo M, Pugliese N, Del Poggio P, Perricone G, Massironi S, Spinetti A, Buscarini E, Vigano M, Carriero C, Fagiuoli S, Aghemo A, Belli LS, Luca M, Pedaci M, Rimondi A, Rumi MG, Invernizzi P, Bonfanti P, Lampertico P. High rates of 30-day mortality in patients with cirrhosis and COVID-19. J Hepatol. 2020 Nov;73(5):1063-1071. doi: 10.1016/j.jhep.2020.06.001. Epub 2020 Jun 9. PMID 32526252
- [Background] Qi X, Wang J, Li X, Wang Z, Liu Y, Yang H, Li X, Shi J, Xiang H, Liu T, Kawada N, Maruyama H, Jiang Z, Wang F, Takehara T, Rockey DC, Sarin SK; COVID-Cirrhosis-CHESS Group. Clinical course of COVID-19 in patients with pre-existing decompensated cirrhosis: initial report from China. Hepatol Int. 2020 Jul;14(4):478-482. doi: 10.1007/s12072-020-10051-z. Epub 2020 May 22. PMID 32440857
- [Background] Moon AM, Webb GJ, Aloman C, Armstrong MJ, Cargill T, Dhanasekaran R, Genesca J, Gill US, James TW, Jones PD, Marshall A, Mells G, Perumalswami PV, Qi X, Su F, Ufere NN, Barnes E, Barritt AS, Marjot T. High mortality rates for SARS-CoV-2 infection in patients with pre-existing chronic liver disease and cirrhosis: Preliminary results from an international registry. J Hepatol. 2020 Sep;73(3):705-708. doi: 10.1016/j.jhep.2020.05.013. Epub 2020 May 21. No abstract available. PMID 32446714
- [Background] Qi X, Liu Y, Wang J, Fallowfield JA, Wang J, Li X, Shi J, Pan H, Zou S, Zhang H, Chen Z, Li F, Luo Y, Mei M, Liu H, Wang Z, Li J, Yang H, Xiang H, Li X, Liu T, Zheng MH, Liu C, Huang Y, Xu D, Li X, Kang N, He Q, Gu Y, Zhang G, Shao C, Liu D, Zhang L, Li X, Kawada N, Jiang Z, Wang F, Xiong B, Takehara T, Rockey DC; COVID-Cirrhosis-CHESS Group. Clinical course and risk factors for mortality of COVID-19 patients with pre-existing cirrhosis: a multicentre cohort study. Gut. 2021 Feb;70(2):433-436. doi: 10.1136/gutjnl-2020-321666. Epub 2020 May 20. No abstract available. PMID 32434831
- [Background] He Q, Zhang G, Gu Y, Wang J, Tang Q, Jiang Z, Shao C, Zhang H, Chen Z, Ma B, Liu D, Xie G, Xu D, Huang Y, Zhang H, Liang M, Huang H, Wang Y, Liu H, Yang J, Pan H, Zou S, Li F, Wang F, Liu C, Wang W, Xiong B, Li X, Liu L, Yang J, Qi X. Clinical Characteristics of COVID-19 Patients With Pre-existing Hepatitis B Virus Infection: A Multicenter Report. Am J Gastroenterol. 2021 Feb 1;116(2):420-421. doi: 10.14309/ajg.0000000000000924. No abstract available. PMID 32925195
- [Background] Cornberg M, Buti M, Eberhardt CS, Grossi PA, Shouval D. EASL position paper on the use of COVID-19 vaccines in patients with chronic liver diseases, hepatobiliary cancer and liver transplant recipients. J Hepatol. 2021 Apr;74(4):944-951. doi: 10.1016/j.jhep.2021.01.032. Epub 2021 Feb 6. PMID 33563499
- [Background] Xia S, Duan K, Zhang Y, Zhao D, Zhang H, Xie Z, Li X, Peng C, Zhang Y, Zhang W, Yang Y, Chen W, Gao X, You W, Wang X, Wang Z, Shi Z, Wang Y, Yang X, Zhang L, Huang L, Wang Q, Lu J, Yang Y, Guo J, Zhou W, Wan X, Wu C, Wang W, Huang S, Du J, Meng Z, Pan A, Yuan Z, Shen S, Guo W, Yang X. Effect of an Inactivated Vaccine Against SARS-CoV-2 on Safety and Immunogenicity Outcomes: Interim Analysis of 2 Randomized Clinical Trials. JAMA. 2020 Sep 8;324(10):951-960. doi: 10.1001/jama.2020.15543. PMID 32789505
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Zhang Y, Zeng G, Pan H, Li C, Hu Y, Chu K, Han W, Chen Z, Tang R, Yin W, Chen X, Hu Y, Liu X, Jiang C, Li J, Yang M, Song Y, Wang X, Gao Q, Zhu F. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine in healthy adults aged 18-59 years: a randomised, double-blind, placebo-controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Feb;21(2):181-192. doi: 10.1016/S1473-3099(20)30843-4. Epub 2020 Nov 17. PMID 33217362